CLINICAL TRIAL: NCT05919537
Title: A Phase 1b Study to Evaluate HMBD-001 With or Without Chemotherapy in Participants With Advanced Solid Tumors Harboring NRG1 Gene Fusions or Selected HER3 Mutations
Brief Title: Study of an Anti-HER3 Antibody, HMBD-001, With or Without Chemotherapy in Patients With Solid Tumors Harboring an NRG1 Fusion or HER3 Mutation
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hummingbird Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMBD-001-102
Record Dates: First submitted 2023-06-01; First posted 2023-06-26 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Non-Small Cell Lung Cancer; Pancreatic Cancer; Locally Advanced Solid Tumor; Metastatic Solid Tumor
Keywords: HMBD-001; NRG1 fusion; NRG1; Neuregulin 1; ErbB3; HER3
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Neoplasm Metastasis; Fibromatosis, Gingival, 2 | interventions — Docetaxel; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A (Experimental): Participants with locally advanced or metastatic pancreatic ductal adenocarcinoma (PDAC) harboring NRG1 gene fusions
  Interventions: Drug: HMBD-001; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Arm B (Experimental): Participants with non-small cell lung cancer (NSCLC) harboring NRG1 gene fusions
  Interventions: Drug: HMBD-001; Drug: Docetaxel
- Arm C (Experimental): Participants with other solid tumors harboring NRG1 gene fusions
  Interventions: Drug: HMBD-001
- Arm D (Experimental): Participants with solid tumors harboring selected HER3 extracellular mutations
  Interventions: Drug: HMBD-001

INTERVENTIONS:
Drug: HMBD-001 — HMBD-001 is a humanized IgG1 anti-HER3 monoclonal antibody (mAb). It is administered IV weekly
Drug: Docetaxel — Docetaxel 75 mg/m^2 IV once every 3 weeks
  Arms: Arm B
Drug: Nab-paclitaxel — Nab-paclitaxel 125 mg/m^2 IV on days 1, 8, 15, every 4 weeks
  Arms: Arm A
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 IV on days 1, 8, 15, every 4 weeks
  Arms: Arm A

SUMMARY:
This is a phase 1b multi-center, open-label study of HMBD-001 with or without chemotherapy in participants with advanced solid tumors harboring NRG1 gene fusions or selected HER3 mutations.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and be willing to sign an informed consent form

  * Males and females aged over 18 years
  * Eastern Cooperative Oncology Group (ECOG) status of 0 to 1
  * Histologic or cytologic evidence of an advanced malignant solid that is resistant/refractory to standard systemic therapy, or for which there is no standard systemic therapy or reasonable therapy in the physician's judgment likely to result in clinical benefit, or the participant has demonstrated to be intolerable to such therapy, or if such therapy has been refused by the participant
  * Arms A, B and C: Cancer harboring an NRG1 gene fusion with EGF-like domain; Arm A: Participants with locally advanced or metastatic pancreatic adenocarcinoma that have not received prior treatment with gemcitabine or nab-paclitaxel and /or have not received more than 2 lines of systemic therapy for advanced disease; Arm B: Participants with locally advanced or metastatic non-small cell lung cancer that have not received prior treatment with docetaxel and /or have not received more than 2 lines of systemic therapy for advanced disease; Arm C: Participants must not be eligible to participate in Arm A or B
  * Arm D: Cancer harboring selected HER3 mutations limited to the extracellular domain.
  * Have an estimated life expectancy of at least 3 months
  * Have an archival tumour sample available or have a site of disease amenable to biopsy and be willing to undergo a biopsy prior to the receipt of the assigned study treatment
  * Have adequate organ function
  * Females must be non-pregnant and non-lactating, willing to use a highly effective method of contraception from screening until study completion or be either surgically sterile or post-menopausal
  * Males must be surgically sterile, abstinent, or if engaged in sexual relations with a woman of child-bearing potential, the participant and his partner must be surgically sterile or using an acceptable, highly effective contraceptive method from screening until study completion

Exclusion Criteria:

* Prior treatment with HMBD-001, pertuzumab, or an agent that specifically targets HER3, including pan-HER tyrosine kinase inhibitors

  * Persistent clinically significant toxicities (Grade ≥2) from previous anti-cancer therapy except for Grade >2 toxicities that are considered unlikely to put the participant at an increased risk of treatment-related toxicity and/or impact the study results e.g., alopecia
  * Most recent anti-cancer therapy including radiotherapy at least 4 weeks, or nitrosourea or mitomycin 3 at least 6 weeks, or 5 half-lives whichever is shorter prior to starting the assigned study treatment
  * Symptomatic primary Central Nervous System (CNS) cancer or metastases unless the symptoms are stable for at least 28 days prior to the first dose of the study drug and any symptoms have returned to baseline
  * Evidence of abnormal cardiac function
  * History of uncontrolled allergic reactions and/or known expected hypersensitivity to the study drugs used in the treatment arm to which the participant is to be enrolled into
  * Any other known active malignancy except for treated cervical intraepithelial neoplasia, or non-melanoma skin cancer
  * Any uncontrolled illness or significant uncontrolled condition(s) requiring systemic treatment
  * Known Human Immunodeficiency Virus (HIV) infection
  * Active hepatitis B or hepatitis C infection
  * Pregnant or breast feeding
  * COVID 19 infection within 3 months prior to the first dose of the study drug
  * COVID 19 vaccination within 14 days prior to the first dose of the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2031-03-01 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and Nature of Adverse Events (AEs) | From the time the ICF is signed until 30 days after last dose of study treatment
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered to be related to the study treatment.
Arm A and B only: Incidence and nature of dose-limiting toxicities (DLTs) during the first cycle of treatment | Arm A: During the first four weeks of study treatment Arm B: During the first three weeks of study treatment
  DLTs will be assessed during the safety run-in phase and are defined as toxicities that meet pre-defined severity criteria and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, intercurrent illness, or concomitant medications that occurs within the first cycle (4 weeks for Arm A, 3 weeks for Arm B) of treatment
Objective Response Rate (ORR) by RECIST V1.1 | Up to 24 months
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - GenesisCare North Shore, Sydney, New South Wales
  - ICON Cancer Centre South Brisbane, Brisbane, Queensland
  - Southern Oncology Clinical Research Unit, Adelaide, South Australia
  - Cabrini Health, Malvern, Victoria
  - Linear Clinical Research, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No